CLINICAL TRIAL: NCT04732806
Title: A Mightier Healthcare System: Introducing a Game-based Pediatric Mental Health Intervention Into Payor-sponsored Care to Evaluate Financial and Clinical Outcomes
Brief Title: A Mightier Healthcare System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neuromotion Labs (Industry)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Magellan Healthcare (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: NML-2020-001; 1R44MH124574-01 (NIH)
Record Dates: First submitted 2021-01-25; First posted 2021-02-01 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Emotional Dysregulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment as usual (No Intervention)
- Intervention (Experimental): Six months of ad lib Mightier play in home
  Interventions: Behavioral: Mightier video games

INTERVENTIONS:
Behavioral: Mightier video games — Biofeedback video game play in home
  Arms: Intervention

SUMMARY:
Access to effective pediatric mental health treatment is a major public health concern in the United States as paucity of pediatric providers leading to long wait times, financial burden, and stigma pose significant barriers to treatment. Digital mental health promises to remedy many chronic problems faced in providing timely and accessible mental health interventions to children. With that in mind, the investigators and Neuromotion Inc. created Mightier, an app-based heart rate biofeedback videogame platform designed to teach and facilitate practice of emotional regulation skills. The technology behind Mightier is backed by three trials showing clinical efficacy and since commercial launch 75% of families who have engaged with the product report improvement. However, Neuromotion's core mission remains increasing access to care, and the direct-to-consumer distribution of digital health also faces access challenges. The investigators propose that access to effective digital mental health interventions can be increased by meeting families where they already know to seek care: the traditional healthcare system. The investigators have partnered with a nationwide behavioral health insurance provider to pilot the integration of Mightier with traditional healthcare. Families will be recruited via direct outreach, social media, or healthcare provider referral. Participating children will be randomized into Mightier or treatment as usual control groups for 6 months. Behavioral healthcare utilization will be observed for 12 months. Through this work the investigators will demonstrate the value of Mightier to various stakeholders via decreased long-term healthcare utilization, confirm that Mightier use results in decreased symptoms of emotional dysregulation, irritability, and parent stress, and explore relationships among Mightier use, healthcare utilization, and symptoms. Ultimately this work will pave the way forward for large scale integration of digital healthcare and more traditional healthcare avenues while simultaneously increasing Mightier's ability to reach children in need.

ELIGIBILITY:
Inclusion:

* Age 8-12
* Insurance provided by Magellan Healthcare OR participant is covered by insurance in Massachusetts and has access to Explanation of Benefits information via online portal
* Has made a behavioral health claim in the past year
* MOAS score of greater than or equal to 2
* Evidence of ADHD, ODD, CD, DMDD, IED, or ASD by MINI-KID
* Parent or guardian is fluent in English
* WiFi at home (for Mightier tablet connection)
* Access to a computer or tablet in the home

Exclusion:

* IQ < 70 (by medical record or clinician judgment)
* Extremely limited verbal capacity
* Change in medication or medication dosage in the past month or planned change in medication or medication dosage in the next month
* Active suicidal ideation
* History of suicide attempt and current depression
* Physical limitations that preclude the use of Mightier
* Sensory sensitivities that would preclude wearing an arm (or leg) heart rate monitor
* Evidence of psychosis, mania, alcohol use disorder, substance use disorder, or PTSD by MINI-Kid
* Ongoing or within the month prior to baseline visit placement in foster care or residential facility

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 183 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2022-11-23 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
Behavioral healthcare utilization cost | 12 Months
  Dollars spent on behavioral healthcare over the study period.
Change in Modified Overt Aggression Scale (MOAS) from baseline to 3 Months | Baseline, 3 months
  The MOAS is a 5-point parent rated scale that rates the severity of four types of aggression: verbal, against property, against self (auto-aggression), and physical towards others. Scores range from 0-100 with lower scores representing less aggression (better outcome).

SECONDARY OUTCOMES:
Change in Disruptive Behavior Disorder Rating Scale (DBDRS) - Oppositional/Defiant Factor Score from baseline to 3 Months | Baseline, 3 months
  The DBDRS is a 45-item scale that evaluates symptoms of Oppositional Defiant Disorder (ODD), Conduct Disorder (CD), and Attention Deficit Hyperactivity Disorder (ADHD) from the parent's perspective. Scores range from 0-135 with lower scores representing fewer behaviors associated with the above disorders (better outcome). This secondary outcome will include the Oppositional/Defiant Factor Score consisting of items 3, 13, 15, 17, 24, 26, 28, and 39.
Change in Affective Reactivity Index - Parent (ARI-P) from baseline to 3 Months | Baseline, 3 months
  The ARI is a 7-item scale that consists of 6 symptom items and 1 impairment item. The scale was designed to determine irritable mood rather than behavioral consequences such as hostility and acts of aggression. Scores range from 0 - 12 with lower scores representing less irritability.
Change in Parent Stress Index - Short Form (PSI-SF) from baseline to 3 Months | Baseline, 3 months
  The PSI-SF is a 36 item parent report scale that evaluates the extent and source of parent stress in the form of three subscales: Parental Distress, Parent-Child Dysfunctional Interaction, and Difficult Child. Total scores range from 36-180 with lower scores representing less parent stress.
Clinical Global Impression - Improvement, Irritability/Anger (CGI-I Irritability/Anger) | 3 months
  The CGI-I scale requires the clinician to rate total improvement whether or not, in the raters judgment, it is due to treatment. The clinician compares the patient's condition at baseline to the time of rating on a scale ranging from 1 (very much improved) to 7 (very much worse)
Clinical Global Impression - Improvement, Aggression (CGI-I Aggression) | 3 months
  The CGI-I scale requires the clinician to rate total improvement whether or not, in the raters judgment, it is due to treatment. The clinician compares the patient's condition at baseline to the time of rating on a scale ranging from 1 (very much improved) to 7 (very much worse)
Clinical Global Impression - Improvement, Oppositional/Defiant Behavior (CGI-I Oppositional/Defiant Behavior) | 3 months
  The CGI-I scale requires the clinician to rate total improvement whether or not, in the raters judgment, it is due to treatment. The clinician compares the patient's condition at baseline to the time of rating on a scale ranging from 1 (very much improved) to 7 (very much worse)
Clinical Global Impression - Improvement, Disruptive Behavior (CGI-I Disruptive Behavior) | 3 months
  The CGI-I scale requires the clinician to rate total improvement whether or not, in the raters judgment, it is due to treatment. The clinician compares the patient's condition at baseline to the time of rating on a scale ranging from 1 (very much improved) to 7 (very much worse)
Change in Parent Confidence and Resources from baseline to 3 Months | Baseline, 3 months
  Two 5 item questions regarding parent confidence in their ability to manage their child's behaviors and adequacy of resources to manage their child's behaviors
Change in NIH-Emotion Toolbox from baseline to 3 Months | Baseline, 3 months
  The NIH toolbox for emotion was developed to create a standardized, comprehensive, and concise battery of tests that can recognize the full spectrum of emotional experiences and their impacts on health and wellbeing. The NIH Toolbox for emotion includes 4 subdomains: negative affect, psychological well-being, stress and self-efficacy, and social relationships. For the age range of 8-12, self-report and proxy measures are available. Given that we expect a wide range of cognitive, developmental, and metacognitive abilities, proxy report measures will be used.

OTHER OUTCOMES:
Customer Satisfaction | 3 months
  Evaluated in the Mightier group only. Customer satisfaction will be rated using a single, parent/guardian response item. Response options will be extremely dissatisfied, somewhat dissatisfied, neither satisfied not dissatisfied, somewhat satisfied, or extremely satisfied.
Net Promoter Score | 3 months
  Evaluated in the Mightier group only. Net Promotor Score represents the industry standard for evaluating customer willingness to recommend a product. The rating consists of a single parent/guardian report item with responses options ranging from 0 (not at all likely) to 10 (extremely likely). When scores are aggregated, Net Promoter Score is expressed as the percentage of customers who rated their likelihood to recommend the product as 9 or 10 minus the percentage of customers rating this at 6 or below.
Heart Rate | 1hz intervals when playing game for 6 months
Change in Disruptive Behavior Disorder Rating Scale (DBDRS) - Total Score | Baseline, 3 Months
  The DBDRS is a 45-item scale that evaluates symptoms of Oppositional Defiant Disorder (ODD), Conduct Disorder (CD), and Attention Deficit Hyperactivity Disorder (ADHD) from the parent's perspective. Scores range from 0-135 with lower scores representing fewer behaviors associated with the above disorders (better outcome).
Behavioral healthcare utilization cost -- billed as medical | 12 Months
  Dollars spent on healthcare billed as medical cost, but related to behavioral or mental health indications, over the study period

CONTACTS AND LOCATIONS:
Locations (1):
- Neuromotion Inc, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No